CLINICAL TRIAL: NCT07206927
Title: Analysis of the Determinants of the Participation of Patients and Health Professionals of the University Hospital Center of Martinique in Clinical Research Protocols in Medical Oncology
Brief Title: Analysis of the Determinants of the Participation of Patients and Health Professionals of the University Hospital Center of Martinique in Clinical Research Protocols in Medical Oncology (StudyOrec)
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital Center of Martinique (Other)
Collaborators: KaFE Association (Karaib Formation Etudes) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 24_RIPH3-04; 2025-A01419-40 (Other: ID-RCB)
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Oncologic Diseases; Cancer; Oncology
Keywords: clinical research participation; investigation; interrogation; barriers and levers of participation; questionnaire
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Qualitative Study : Patients interviews: For the qualitative part, 30 patients will be included in the study. A semi-structured interview, lasting 20 to 30 minutes, will be conducted by the sociologist and anthropologist. They will use questionnaires (semi-structured interview grids), administered to patients face-to-face or by telephone. Patients will be interviewed only once.
  The interview grid includes the following sections: personal characteristics such as age, family and professional situation, municipality of residence, and knowledge of clinical research.
  Interventions: Other: Qualitative Study: Semi-structured interview for patients
- Quantitative Study : Healthcare professionals questionnaires: For the qualitative part, 30 healthcare professionnals will be included in the study.
  Questionnaires will be administered by email, in a single session, to healthcare professionals who have agreed to participate in the study.
  Interventions: Other: Quantitative Study : Healthcare professionals questionnaires

INTERVENTIONS:
Other: Qualitative Study: Semi-structured interview for patients — A semi-structured interview, lasting 20 to 30 minutes, will be conducted by the sociologist and anthropologist. They will use questionnaires (semi-structured interview grids), administered to patients face-to-face or by telephone. Patients will be interviewed only once. The interview grid includes the following sections: personal characteristics such as age, family and professional situation, municipality of residence, and knowledge of clinical research.
  Groups: Qualitative Study : Patients interviews
Other: Quantitative Study : Healthcare professionals questionnaires — Questionnaires will be administered by email, in a single session, to healthcare professionals who have agreed to participate in the study.
  Groups: Quantitative Study : Healthcare professionals questionnaires

SUMMARY:
For optimal patient care, it is imperative that healthcare professionals implement appropriate strategies. These strategies must take into account changes in healthcare practices associated with advances in medications and medical equipment. Clinical trials play a crucial role in validating the efficacy and safety of these advances, ensuring high-quality and constantly improving healthcare.

However the proportion of patients included in therapeutic trials is often considered too low.

Several ideas have been explored to explain the low participation rate in research projects. These are closely linked to research actors and tools, such as, for example:

* the research protocol and its eligibility criteria, which may be overly strict
* healthcare professionals with the barriers encountered in carrying out research programs (motivation, attitude and perceptions, human, logistical and technical constraints, lack of training)
* patients who are generally poorly acculturated to clinical research, the lack of information for patients in healthcare services, and patients' lack of trust in the healthcare system.
* ...

In Martinique, healthcare professionals face the same challenges in including patients in clinical trials.

Patient inclusion is necessary due to the region's demographic and medical characteristics. To improve patient inclusion in these trials, it is important to define the human and material barriers and levers that influence the participation of patients and healthcare professionals in clinical research protocols in the medical oncology departments of the Martinique University Hospital.

The investigators believe that increased patient awareness of the benefits of clinical research, equally increased incentives for healthcare professionals, and the establishment of adequate support structures would increase participation in clinical research protocols within the medical oncology departments of the Martinique University Hospital.

By conducting a mixed qualitative and quantitative study to gather the perspectives of patients and caregivers, the investigators aim to identify the human and material barriers that limit the participation of oncology patients in Martinique.

DETAILED DESCRIPTION:
As the French department with the oldest population, Martinique faces an over-incidence of certain diseases. For optimal patient care, it is imperative that healthcare professionals implement appropriate strategies. These strategies must take into account changes in healthcare practices associated with advances in medications and medical equipment. Clinical trials play a crucial role in validating the efficacy and safety of these advances, ensuring high-quality and constantly improving healthcare.

The goal of clinical research is to improve knowledge about a medication, a pathology, a procedure, or a treatment protocol.

Regardless of the specialty, clinical trials remain the only scientific means of demonstrating the quality and accuracy of information or the safety of medications or medical techniques.

Furthermore, offering a patient the opportunity to participate in a clinical trial is often a source of therapeutic alternatives or innovations.

It should be noted that the proportion of patients included in therapeutic trials is often considered too low.

Several ideas have been explored to explain the low participation rate in research projects. These are closely linked to the research stakeholders and tools. These include:

* The research protocol, particularly the eligibility criteria: In a survey conducted among sponsors on the factors influencing recruitment, the major barrier cited was identifying subjects who meet the eligibility criteria. These can be very strict, limiting the number of eligible patients.
* Healthcare professionals with the barriers encountered in carrying out research programs: They may be related to the investigator themselves (their motivation, attitude, and perceptions).

These parameters can have an impact on the patient's choice. In this study, the authors highlight the importance played by the investigator in recommending the trial to the patient. This is a decisive factor in their decision to participate in a clinical trial. This clearly demonstrates the trust patients place in their physician as the primary source of information regarding clinical trials.

There may also be limitations in terms of human, logistical, and technical constraints. Indeed, a lack of human resources is a recurring problem in research centers. Thus, after eligibility criteria, the second obstacle to patient participation in research projects is the lack of human resources at centers for patient recruitment (67% of respondents). Physicians are already overworked with care and may lack both logistical support and time to assist with recruitment.

A lack of training and specialized staff, as well as physicians' fear of negative reactions from their patients and the risk of disrupting the doctor-patient relationship of trust, are all factors also addressed in these articles.

* Patients with a lack of information: Few patients (15%) report being informed about ongoing clinical trials, while a greater number (75%) express a positive desire to participate in a clinical trial if they were aware of them. Patients may also not understand the importance of clinical trials or have concerns about the safety of clinical trials, the side effects of experimental treatments, or the possibility of receiving a placebo rather than the active treatment. There is also the trust that patients may place in the research world. Some patients may lack trust in the medical research system, which may discourage them from participating in clinical trials.
* Selection of trial sites: Clinical trials may not be available in all regions. Indeed, in their study by Allignet et al. show that the density of clinical trials in the French overseas departments is significantly lower than in mainland France, except in onco-dermatology.

Other authors have explored cross-cutting themes such as the association between scientific production and a specific research area or the inclusion of patients from ethnic and racial minorities in clinical trials.

In Martinique, healthcare professionals face the same challenges in including patients in clinical trials.

Patient inclusion is necessary due to the region's demographic and medical characteristics. To improve patient inclusion in these trials, it is important to define the human and material barriers and levers that influence the participation of patients and healthcare professionals in clinical research protocols in the medical oncology departments of the Martinique University Hospital.

Research Hypotheses:

The investigators believe that increased patient awareness of the benefits of clinical research, equally increased incentives for healthcare professionals, and the establishment of adequate support structures would increase participation in clinical research protocols within the medical oncology departments of the Martinique University Hospital.

By conducting a mixed qualitative and quantitative study to gather the perspectives of patients and caregivers, the investigators aim to identify the human and material barriers that limit the participation of oncology patients in Martinique.

The qualitative method requires the support of professionals in the humanities and social sciences (HSS) who can provide methodological support and experience in patient interviews.

This is why the research team chose to be accompanied by a sociologist and an anthropologist who already have experience in the health field in Martinique, particularly with patients suffering from prostate cancer.

Secondly, the results of this study will be used to establish appropriate organizational structures for the participation of patients in Martinique in oncology clinical research protocols.

ELIGIBILITY:
Inclusion Criteria for patients group:

* Male or female,
* Age ≥ 18 years,
* Patient being treated for cancer at the University Hospital Center of Martinique,
* Patient who can read and/or understand French,
* Patient who has consented to the use of their medical data for this research.

Inclusion Criteria for professionals group:

- Any qualified healthcare professional working in the medical oncology departments of the University Hospital Center of Martinique, such as oncologists, radiation therapists, urologists, nurses, etc.

Exclusion Criteria for patients group:

* Patient with known cognitive impairments that prevent them from completing the questionnaire,
* Subjects under legal protection (guardianship/curatorship),
* Subjects at an advanced stage of the disease (asthenia),
* Written or oral objection from the patient to the use of data for research purposes.

Exclusion Criteria for professionals group:

* Students in training regardless of their field,
* Replacement healthcare professionals for a period of less than 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: * Patient being treated for cancer at the University Hospital Center of Martinique.
  * Qualified healthcare professional working in the medical oncology departments of the University Hospital Center of Martinique.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative study with patients: questioning the participation of patients from the services involved in medical oncology at the Martinique University Hospital in clinical research projects and identifying the obstacles and levers to this participation. | 6 months
  A semi-structured interview, lasting 20 to 30 minutes, will be conducted by the sociologist and anthropologist. They will use questionnaires (semi-structured interview grids), administered to patients face-to-face or by telephone. Patients will be interviewed only once. The interview grid includes the following sections: personal characteristics such as age, family and professional situation, municipality of residence, and knowledge of clinical research.
Quantitative study among professionals: measure the proportion of healthcare professionals of CHU of Martinique who have already participated in clinical research projects or agreed to participate in them treating patients with medical oncology needs. | 3 months
  Questionnaires will be administered by email, in a single session, to healthcare professionals who have agreed to participate in the study.

SECONDARY OUTCOMES:
Qualitative patient study: Research the existence of factors associated with patient participation such as age, gender, socio-professional category, etc. | 6 months
  Factors such as age, gender, socio-professional category, etc... will be studied.
Quantitative study among professionals: Measure the importance of identified barriers and enablers for participating in clinical research projects among healthcare professionals in the medical oncology departments of the Martinique University Hospital. | 3 months
  Percentages obtained for each lever or brake identified.

CONTACTS AND LOCATIONS:
Overall Officials: Mickaëlle ROSE, Principal Investigator — University Hospital Center of Martinique
Locations (1):
- University Hospital Center of Martinique, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No